CLINICAL TRIAL: NCT04303650
Title: The Relation Between Sonographic Quadriceps Muscle Layer Thickness and Nitrogen Balance for Nutrition Monitoring in Adult Critically Ill Trauma Patients
Brief Title: The Relation Between Quadriceps Muscle Layer Thickness and Nitrogen Balance for Nutrition Monitoring
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sherif M. S. Mowafy, Lecturer of anesthesia and surgical intensive care, Zagazig University
Other Study IDs: 5968-5-3-2020
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound measurement of quadriceps muscle layer thickness — With patient in supine position ultrasound will be performed using a 12MHZ Transducer connected to Sonosite M Turbo machine. The probe will be placed perpendicular to the long axis of the thigh on its anterior surface at the two thirds of the length between the anterior superior iliac spine and the upper border of the patella. After identifying the muscle tissue, the thickness of the quadriceps muscle will be obtained by measuring the distance between the cortex of femur and the most superficial muscular fascia. Measurements will be performed by applying maximal compression on the probe without inflicting pain to prevent underestimation of muscle wasting linked to subcutaneous edema. measurements will be made on both sides repeatedly on ICU days 1, 3, 7, and 10. Every time three ultrasound measurements will be taken per site and the average of three measurements for each site will be used and combined to provide total muscle depth

SUMMARY:
Loss of muscle mass is a major cause of intensive care unit-acquired weakness (ICU-AW) and is associated with delayed weaning; prolonged ICU and hospital stay and is an independent predictor of one year mortality.

Theoretically, the best strategy to minimize muscle loss during ICU stay, is delivering an appropriate nutritional support. Studying the correlation between the sequential assessments of quadriceps femoris muscle layer thickness (QMLT) by the aid of Ultrasound in addition to the traditional method (NB) for assessment of nutritional status may be helpful to predict outcome and mortality.

DETAILED DESCRIPTION:
Protein catabolism and proteolysis, mainly in the skeletal muscles is highly accelerated in critical illness with severe acute inflammatory processes, such as sepsis, burns, and polytrauma patients. The resulting catabolic state may be linked to immunosuppression, poor wound healing, and intensive care unit-acquired weakness (ICU-AW), which are associated with delayed recovery and increased mortality. In order to prevent muscle-protein depletion, several strategies have been proposed. One of them is adequate nutrition. Higher protein intake appears to be beneficial and could mitigate the negative catabolic state by increasing the availability of exogenous amino acids.

The adequacy of protein intake could only be optimized by appropriate monitoring. Nitrogen balance (NB) is the commonly used tool in this context. It is considered a good marker of adequate protein intake, easy, and available method of assessing the success of nutritional therapy as it reflects the gain or loss of total body proteins by calculating the difference between dietary nitrogen intake and nitrogen losses.

Moreover, a considerable reduction in muscle mass begins within the first 3 days of ICU admission and progressively worsens; therefore quantifying the muscle size may help in recognizing patients at risk of ICU acquired weakness and also may guide the interventions to prevent this complication. So, it may help in monitoring the adequacy of nutritional therapy and protein intake.

The primary methods that have been explored to measure musculature include computed tomography (C.T), magnetic resonance imagining (MRI), ultrasonography (US), and bioimpedance. Ultrasonography as a noninvasive, practical, readily available, and bedside technique could be considered the first option for the quantification of muscle size in these patients.

The quadriceps muscle is the most studied muscle found to have strong correlation with muscle mass and strength. Its size can be measured by either the quadriceps muscle layer thickness (QMLT) or the cross-sectional area (CSA). However, QMLT have greater practicability as measurements could be obtained rapidly and in real time as well as it easier to identify than CSA.

Since, monitoring is the key to individualize and optimize the critical protein intake. We hypothesized that QMLT evaluation by ultrasound could be used to guide nutritional protein intake and is correlated to conventional monitoring with nitrogen balance in critically ill trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated to be mechanically ventilated to >48hour and expected to Stay in ICU > 4 days.
* No contraindication to early enteral nutrition.
* Enteral feeding in the first 24 hours after admission, with a minimum protein contribution of 1 gm / kg / day.
* We recruited only well nourished, previously healthy patients with no past history of nutritional problems.

Exclusion Criteria:

* Patients with preexisting neuromuscular pathology, lower limb amputation, skeletal fractures or immobilization in the previous 2years.
* Patients with relevant Co-morbidities (renal, liver or heart disease or COPD), previous immune abnormalities including those receiving corticosteroids, and those with past or recent history of cancer.
* Patients with anuria owing to the difficulty in evaluating excreted urea nitrogen
* Whose ultrasound data will be missing or incomplete
* Pregnancy
* Patients who will not reach the goal in enteral protein intake for any reason (gastrointestinal intolerance, contraindication to enteral feeding or repeated interruptions of enteral feeding due to multiple surgical procedures) or those who start parenteral nutrition.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Critically ill trauma patients aged between 18 - 60 years of both sexes
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
correlation between Nitrogen Balance and quadriceps muscle layer thickness (QMLT) | 10 days
  To determine the correlation between Nitrogen Balance and QMLT detected by ultrasound

SECONDARY OUTCOMES:
relationship between QMLT, pre-albumin, and CRP | 10 days
  To determine the correlation between pre-albumin and CRP and QMLT detected by ultrasound
The impact of QMLT and NB on 28 day mortality. | 28 day
  To determine the correlation between nitrogen balance and QMLT detected by ultrasound and the outcome by 28 day mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma M Ahmed, MD, Study Director — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University; Sherif MS Mowafy, MD, Principal Investigator — Anesthesia and Surgical Intensive Care Department, Faculty of Medicine, Zagazig University
Locations (1):
- Emergency and Surgical Intensive Care Units, Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the IPD and any additional supporting information will become available starting 6 months after publication.
Access Criteria: by contacting the study director

REFERENCES:
- [Background] Liebau F, Wernerman J, van Loon LJ, Rooyackers O. Effect of initiating enteral protein feeding on whole-body protein turnover in critically ill patients. Am J Clin Nutr. 2015 Mar;101(3):549-57. doi: 10.3945/ajcn.114.091934. Epub 2015 Feb 4. PMID 25733640
- [Background] Fock RA, Blatt SL, Beutler B, Pereira J, Tsujita M, de Barros FE, Borelli P. Study of lymphocyte subpopulations in bone marrow in a model of protein-energy malnutrition. Nutrition. 2010 Oct;26(10):1021-8. doi: 10.1016/j.nut.2009.08.026. Epub 2009 Dec 29. PMID 20036516
- [Background] Rai J, Gill SS, Kumar BR. The influence of preoperative nutritional status in wound healing after replacement arthroplasty. Orthopedics. 2002 Apr;25(4):417-21. doi: 10.3928/0147-7447-20020401-17. PMID 12002213
- [Background] Latronico N, Herridge M, Hopkins RO, Angus D, Hart N, Hermans G, Iwashyna T, Arabi Y, Citerio G, Ely EW, Hall J, Mehta S, Puntillo K, Van den Hoeven J, Wunsch H, Cook D, Dos Santos C, Rubenfeld G, Vincent JL, Van den Berghe G, Azoulay E, Needham DM. The ICM research agenda on intensive care unit-acquired weakness. Intensive Care Med. 2017 Sep;43(9):1270-1281. doi: 10.1007/s00134-017-4757-5. Epub 2017 Mar 13. PMID 28289812
- [Background] Andonovska, B.J., Andonovski, A.G., Kuzmanovska, B., Kartalov, A., Temelkovski, Z. the influence of nutrition on muscle wasting in critically ill patients - a pilot study.Sanamed 2018; 13(3):235 - 41
- [Background] Felicetti-Lordani CR, Eckert RG, Valerio NMP,et al. Nitrogen balance in nutritional monitoring of critically ill adult patients:A prospective observational study.Yoğun Bakım Derg 2018; 8: 59-64.
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Nakanishi N, Oto J, Tsutsumi R, Iuchi M, Onodera M, Nishimura M. Upper and lower limb muscle atrophy in critically ill patients: an observational ultrasonography study. Intensive Care Med. 2018 Feb;44(2):263-264. doi: 10.1007/s00134-017-4975-x. Epub 2017 Nov 6. No abstract available. PMID 29110031
- [Background] Price KL, Earthman CP. Update on body composition tools in clinical settings: computed tomography, ultrasound, and bioimpedance applications for assessment and monitoring. Eur J Clin Nutr. 2019 Feb;73(2):187-193. doi: 10.1038/s41430-018-0360-2. Epub 2018 Oct 30. PMID 30377307
- [Background] Weinel LM, Summers MJ, Chapple LA. Ultrasonography to measure quadriceps muscle in critically ill patients: A literature review of reported methodologies. Anaesth Intensive Care. 2019 Sep;47(5):423-434. doi: 10.1177/0310057X19875152. Epub 2019 Oct 22. No abstract available. PMID 31640395
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Background] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463